CLINICAL TRIAL: NCT06441305
Title: Assessing the Impact, Implementation and Cost of Empowering Community Health Promoters to Improve Wasting Treatment Coverage in Turkana County Through Family-led MUAC Scale-up, Weight-for-age Screening, and Defaulters' Follow-up
Brief Title: Expanding Coverage of Severe Acute Malnutrition (SAM) Treatment in Kenya
Acronym: R-SWITCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: UNICEF (Other); Kenyatta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RSWITCH-Kenya
Record Dates: First submitted 2024-05-06; First posted 2024-06-04 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Acute Malnutrition, Severe; Malnutrition, Child; Wasting
Keywords: Outpatient Therapeutic Feeding Program; Treatment; Screening; Wasting; Severe acute malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition; Child Nutrition Disorders; Cachexia

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial. Unit/cluster of assignment is community unit catchment area. Parallel Assignment: baseline-endline design
Masking Description: Evaluator teams will be blinded from intervention allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): * Register-based household registration (census) by CHP every 12 months
  * Some family MUAC of variable and unknown coverage/frequency, national guidance developed.
  * Some passive screening using weight-for-height z-score at Health Facility and during outreach during Malezi bora (child health week every 6 months).
  * Monthly compilation by CHA (supervisors) of the list of defaulters and non-respondents for transmission to relevant community health promoter (CHP) during monthly in-person meeting.
- SWITCH intervention package (Experimental): * Addition of digital monitoring & supervision by CHA
  * Digitized registration of households by CHPs every 6 months
  * Digital reminders to CHP to conduct home visit if a child has never been visited in 3 mo.
  * Digital reminder for timely training to family MUAC of all family members through home visit by CHP when child turns 6 months of age.
  * Platform for 2-ways messaging: biweekly SMS reminders to caregivers through the CHP's app; feedback by caregiver
  * Community level screening based on weight and weight-for-age (WAZ) led by CHP every other month (aligned with Community Action Days),
  * Digital calculation of WAZ.
  * CHP and Growth Monitoring and Promotion refer to health facility if WAZ<-3 to check on WHZ eligibility
  * At the end of every wasting treatment consultation, compilation of the list of defaulters and non-respondents, for immediate transmission by CHA to relevant CHP through digital task of an instruction for immediate follow-up.
  Interventions: Behavioral: SWITCH intervention package

INTERVENTIONS:
Behavioral: SWITCH intervention package — * Addition of digital monitoring & supervision by CHA
  * Digitized registration of households by CHPs every 6 months
  * Digital reminders to CHP to conduct home visit if a child has never been visited in 3 mo.
  * Digital reminder for timely training to family MUAC of all family members through home visit by CHP when child turns 6 months of age.
  * Platform for 2-ways messaging: biweekly SMS reminders to caregivers through the CHP's app; feedback by caregiver
  * Community level screening based on weight and weight-for-age (WAZ) led by CHP every other month (aligned with Community Action Days),
  * Digital calculation of WAZ.
  * CHP and Growth Monitoring and Promotion refer to health facility if WAZ<-3 to check on WHZ eligibility
  * At the end of every wasting treatment consultation, compilation of the list of defaulters and non-respondents, for immediate transmission by CHA to relevant CHP through digital task of an instruction for immediate follow-up.
  Arms: SWITCH intervention package

SUMMARY:
Child wasting is a type of malnutrition which occurs when a child becomes too thin. This medical condition increases the risk of becoming sick or dying. A child with severe wasting needs to be seen in a medical consultation to check on health status and to receive some medicine and a medical food supplement for daily consumption until cured. Yet, only a small proportion of children suffering from severe wasting are presently receiving appropriate treatment.

In Kenya, there is an opportunity to build on the existing network of community health promoters (CHPs) to increase the number of children with wasting who are identified and treated. In intervention areas, CHPs will be equipped with smartphones and an application which provides guidance on household members to visit and simple actions to take, related to health. CHPs will distribute color-coded mid-upper arm circumference tapes to households with young children and train caregivers on how to use it. After training, CHPs will send Short Message Services (SMS) to remind caregivers to regularly measure the arm circumference of the child. In addition, CHPs will receive a scale to measure the weight of children every month. Finally, wasted children registered in the treatment program who fail to attend a planned consultation will be flagged to their CHP through the phone application, and CHPs will conduct a specific home visit to investigate and help solve potential issues.

The study will assess whether this community intervention (called SWITCH) allows to identify and treat more children suffering from severe wasting. Before the start of the intervention, the proportion of wasted children receiving treatment in 40 community units in Turkana South, Turkana East and Aroo will be assessed. After this survey, a computer will randomly select 20 community units where the intervention will be scaled up. The survey will be repeated after 2 years to assess if the proportion of severely wasted children receiving treatment is higher in the area where the intervention was scaled up compared to the area where it was not scaled up.

In addition, after 1 year of implementation, the study will assess how the intervention was scaled up, what are the main challenges, and what are the overall perceptions on the intervention in the community among those who receive it and those who deliver it. Finally, costs of the various components of the intervention will be measured for all actors involved, including for caregivers.

DETAILED DESCRIPTION:
Despite the burden and impact of child wasting on morbidity and mortality, only a small proportion of severely wasted children are presently receiving treatment. In Kenya, there is an opportunity to strengthen the screening for wasting and the identification and treatment of wasted children (SWITCH) through community health promoters (CHPs) who, per policy, are trained, equipped, incentivized and supervised by community health agents (CHAs).

An intervention package will be implemented including: 1) Digitization to support CHPs, 2) Family-led Mid-Upper Arm Circumference (MUAC) enhanced by digitization, with a two-way messaging platform between CHP and caregivers, and reminders for timely training at 6 months of age, 3) Equipment of CHPs with a baby-mother scale for measurement of weight-for-age to detect likely wasting, and 4) Real-time follow-up in the community (facilitated by digitization) of defaulters and non-respondent children enrolled for wasting treatment.

A randomized controlled trial will be used to assess the impact of the SWITCH intervention on severe wasting treatment coverage in Turkana. Twenty randomly selected community units of 40 will receive the intervention. An exhaustive screening campaign conducted at baseline and endline (after 2 years) in the 40 community units will identify children with severe wasting (MUAC < 115 mm or Weight-for-Height Z-score < -3 or bilateral pitting oedema) or recovering from severe wasting (defined by receipt and consumption of Ready-to-Use Therapeutic Food), who will be enrolled in a survey assessing treatment coverage, program exposure and other pathways to impact, and confounders.

In addition, the study will assess the reach, adoption by CHPs, and implementation challenges of the SWITCH package through additional qualitative (interviews and observations) and quantitative data collection at all levels of program delivery (beneficiaries, CHPs, CHAs, program implementers); and the unit cost of the SWITCH package per beneficiary (and cost-effectiveness if the package is effective) through an activity-based costing-ingredients approach.

ELIGIBILITY:
Inclusion Criteria:

* Household in a village of the study area covered by a CHP (although the child may or may not be registered by a CHP) AND
* Child is 6-59.9 months of age AND
* Caregiver consents to be part of the study AND
* any of the following:

  * WHZ < -3 (relative to WHO 2006 reference) OR
  * MUAC <115 mm OR
  * Presence of bilateral edema OR
  * receiving treatment as follow-up for an initial SAM condition on the way to full recovery

exclusion criteria is:

* Congenital malformation that makes anthropometric measurements impossible.
* Length is below 54 cm or height is above 120cm.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1600 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Period prevalence of severe wasting (SAM) treatment coverage in children 6-59 months of age | After 24 months of program implementation
  defined as the proportion of children suffering from SAM or recovering from SAM who currently receive treatment.
  • SAM defined by weight-for-height Z-score (WHZ) <-3 (relative to World Health Organization (WHO) 2006 reference) or MUAC <115 mm or by the presence of bilateral edema.
  Children recovering from SAM through treatment will be considered to receive treatment for an initial SAM condition if they both attended an IMAM consultation in the previous 15 days (as reported by caregiver OR by a consultation card) AND either:
  * consumed RUTF at least once in the previous 3 days (as reported by the caregiver AND confirmed by observation of >= 1 full or 2 empty RUTF sachets) OR
  * consumed RUSF at least once in the previous 3 days (as reported by the caregiver AND confirmed by observation by the enumerator of >= 1 full or 2 empty RUSF sachets) AND child was previously enrolled for SAM treatment immediately prior to MAM treatment (as confirmed by treatment card OR reported by the mother

SECONDARY OUTCOMES:
Point prevalence of SAM outpatient therapeutic program (OTP) treatment coverage in children 6-59 months of age | After 24 months of program implementation
  Defined as the proportion of children with SAM at the time of the survey that are under treatment (see definition under primary outcome)
Screening coverage of SAM | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months suffering from SAM ((currently or on their way to recovery from SAM through treatment for an initial SAM condition) ) screened for wasting over the last 30 days (as reported by the caregiver)
Prevalence of SAM | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with SAM (defined as WHZ <-3 (relative to World Health Organization (WHO) 2006 reference) or a MUAC < 115 mm or the presence of bilateral pitting edema).
Prevalence of very low WHZ | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with WHZ <-3 (relative to World Health Organization (WHO) 2006 reference).
Prevalence of very low MUAC | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with MUAC<115 mm
Prevalence of moderate acute malnutrition (MAM) | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with MAM (defined as -3<= WHZ <-2 (relative to World Health Organization (WHO) 2006 reference) or 115<= MUAC < 125 mm).
Prevalence of wasting | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months with wasting (defined as WHZ <-2 (relative to World Health Organization (WHO) 2006 reference) or a MUAC < 125 mm or the presence of bilateral pitting edema).
Prevalence of stunting | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months suffering from SAM or recovering from SAM with stunting (defined as height-for-age Z-scores (HAZ) <-2 or a MUAC < 125 mm or the presence of bilateral pitting edema). To calculate HAZ scores the 2006 WHO growth reference will be used
Prevalence of underweight and severe underweight | After 24 months of program implementation
  Defined as the proportion of children aged 6-59 months suffering from SAM or recovering from SAM with underweight (defined as weight-for-age Z-scores (WAZ) <-2 ) and severe underweight (defined as WAZ <-3 ). To calculate WAZ scores the 2006 WHO growth reference will be used
Mean height-for-age Z-score (HAZ) | After 24 months of program implementation
  In 6-59 months old children suffering from SAM or recovering from SAM. Scores will be calculated relative to World Health Organization (WHO) 2006 reference, with a higher score meaning a better outcome
Mean weight-for-height Z-score (WHZ) | After 24 months of program implementation
  In 6-59 months old children.To calculate WHZ scores the 2006 WHO growth reference will be used
Mean weight-for-age Z-score (WAZ) | After 24 months of program implementation
  In 6-59 months old children.To calculate WAZ scores the 2006 WHO growth reference will be used
Mean mid-upper arm circumference (MUAC) | After 24 months of program implementation
  In 6-59 months old children.
Caregiver's knowledge score | After 24 months of program implementation
  The score will be calculated by adding one point for each right answer to a series of questions related to infant and child feeding, child health and hygiene, the condition of severe acute malnutrition, outpatient therapeutic programs, screening of wasting. Questions were specifically developed for the study based on program activities and asked to caregiver of children aged 6-59 months suffering from SAM or recovering from SAM
Prevalence of appropriate immunization | After 24 months of program implementation
  Proportion of children aged 6-18 months with SAM or enrolled in SAM OTP who received all recommended immunizations
Coverage of the integrated management of acute malnutrition (IMAM) platform | After 24 months of program implementation
  proportion of children aged 6-59 months suffering from SAM or recovering from SAM who attended an IMAM consultation in the previous 15 days (as reported by the caregiver or by an IMAM treatment card)
Coverage of the community unit platform | After 24 months of program implementation
  proportion of children aged 6-59 months suffering from SAM or recovering from SAM in contact with a CHP in the 2 months preceding the survey for community care-related matter (as reported by the caregiver)
Coverage of family MUAC | After 24 months of program implementation
  proportion of children aged 6-59 months suffering from SAM or recovering from SAM screened in the month preceding the survey by a family member using a MUAC tape (as reported by the caregiver)
Coverage of family MUAC training | After 24 months of program implementation
  proportion of children aged 6-59 months suffering from SAM or recovering from SAM for which at least one family member was trained to use MUAC tape (as reported by the caregiver)
Coverage of MUAC tapes | After 24 months of program implementation
  proportion of children aged 6-59 months suffering from SAM or recovering from SAM for which at least one family member owns a MUAC tape (as reported by the caregiver AND confirmed by observation)
Coverage of WAZ screening | After 24 months of program implementation
  proportion of children aged 6-59 months suffering from SAM or recovering from SAM weighed in the 2 months preceding the survey by a CHP or a health staff using a scale (as reported by the caregiver)
Mean longitudinal prevalence of child morbidity | After 24 months of program implementation
  In children aged 6-59 months suffering from SAM or recovering from SAM, defined as the number of days of illness (acute respiratory infections, fever, diarrhea, vomiting) in the past 3 days (as reported by the caregiver) divided by the total number of days of report (usually 3). A diarrheal episode is defined as at least three loose stools in the last 24 hours, or stools with blood. Fever will be measured by a thermometer by enumerators and the history of fever in the previous days will also be recalled from the mother. The presence of an acute respiratory infection (ARI) will be assessed by recalling the specific symptoms associated with ARI (cough, difficulty breathing, rapid breathing, runny nose).

CONTACTS AND LOCATIONS:
Overall Officials: Elodie Becquey, PhD, Principal Investigator — International Food Policy Research Institute; Sophie Ochola, PhD, Principal Investigator — Kenyatta University
Locations (1):
- Turkana South and Turkana East and Aroo, Lodwar, Kenya

IPD SHARING:
Plan to Share IPD: Yes
All data will be carefully anonymized and de-identified so that the privacy of participants and research subjects is fully protected. Databases will be anonymized using identification codes. No names, GPS coordinates, dates of birth or other identifying data will be stored in the databases.
  At the time of publication of scientific articles presenting primary results, the fully anonymized databases (quantitative data) will become a public good and will be made available to the scientific community, government, and partners.
Supporting Information: Study Protocol, SAP
Time Frame: At the time of publication of scientific articles presenting primary results.